CLINICAL TRIAL: NCT03660176
Title: Effects of Butyrate Enemas on Postoperative Intestinal Mobility Disorders in Hirschsprung's
Brief Title: Effects of Butyrate Enemas on Postoperative Intestinal Mobility Disorders in Hirschsprung's Disease
Acronym: Buty-Hirsch
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-02
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-08

CONDITIONS: Hirschsprung's Disease
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine management (Active Comparator): Children in the control group receive no additional treatment
  Interventions: Other: routine management
- EXP GROUP (Experimental): children receiving butyrate enemas + routine management butyrate enemas every day before Curative surgery
  Interventions: Drug: butyrate enemas + routine management

INTERVENTIONS:
Drug: butyrate enemas + routine management — 10ml/kg volume of butyrate enemas in addition to the colonic irrigations
  Arms: EXP GROUP
Other: routine management — the colonic irrigations
  Arms: routine management

SUMMARY:
Hirschsprung's disease (HD) is a rare disease defined as a congenital absence of enteric ganglia, resulting usually in neonatal bowel obstruction. The current treatment is the operative removal of the aganglionic bowel and anastomosis to the ganglionic zone considered as 'healthy'. However, postoperative course remains unpredictable.

Functional intestinal disorders are present in up to 45% of patients and can occur in the immediate postoperative period or few weeks/years later.

Until now, there are neither predictive factors of postoperative digestive complications nor established treatment for postoperative dysmotility in HD. Abnormalities in enteric nervous system (ENS) phenotype and functions in the 'healthy' ganglionic segment are increasingly suspected to be directly responsible for postoperative intestinal dysfunctions in HD. Therefore, approaches aimed at restoring the nitrergic phenotype could be of major therapeutical interest. Among targets regulating the nitrergic phenotype of ENS are the microbiota and/or derived metabolites. Indeed preclinical animal models deficient in bacterial sensing molecules have a loss of nitrergic neurons and reduced colonic transit. Conversely, microbiota transfer to newborn germ-free mice restored colonic transit time. Alternatively the investigators has shown that bacterial metabolites such as short-chain fatty acids, in particular butyrate, can increase nitrergic phenotype and enhance colonic motility in a gut immaturity animal model. Therefore the investigators hypothesize preoperative butyrate enema will reduce postoperative intestinal complications at short-term and medium/long-term.

DETAILED DESCRIPTION:
Hirschsprung's disease (HD) is a rare disease (1/5000) defined as a congenital absence of enteric ganglia, secondary to developmental defects in colonization of the gut by the enteric nervous system (ENS) and in its maturation, resulting usually in neonatal bowel obstruction. The current treatment is the operative removal of the aganglionic bowel and anastomosis to the ganglionic zone considered as 'healthy'. However, postoperative course remains unpredictable. Functional intestinal disorders, mainly functional obstructive symptoms, are present in up to 45% of patients and can occur in the immediate postoperative period or few weeks/years later. Postoperative enterocolitis also occurs in up to 25% of patients following a similar time course. Until now, there are neither predictive factors of postoperative digestive complications nor established treatment for postoperative dysmotility in HD, in part due to a lack of understanding of the physiopathological mechanisms involved. Abnormalities in ENS phenotype and functions in the 'healthy' ganglionic segment are increasingly suspected to be directly responsible for postoperative intestinal dysfunctions in HD. In an ongoing multicentre study (Ente-Hirsch project), he investigators have identified a reduced density of nitrergic enteric neurons associated with a reduced neuromuscular transmission that could account for digestive dysfunctions in HD. Therefore, approaches aimed at restoring the nitrergic phenotype could be of major therapeutical interest. Among targets regulating the nitrergic phenotype of ENS are the microbiota and/or derived metabolites. Indeed preclinical animal models deficient in bacterial sensing molecules have a loss of nitrergic neurons and reduced colonic transit. Conversely, microbiota transfer to newborn germ-free mice restored colonic transit time. Alternatively he investigators has shown that bacterial metabolites such as short-chain fatty acids, in particular butyrate, can increase nitrergic phenotype and enhance colonic motility in a gut immaturity animal model. Therefore the investigators hypothesize preoperative butyrate enema will reduce postoperative intestinal complications at short-term and medium/long-term.

ELIGIBILITY:
Inclusion Criteria:

* Newborn with a diagnosis of Hirschsprung's disease the 2 first months of life,
* Born at or after 35 weeks of gestation (37 weeks of amenorrhea),
* With a short-segment Hirschsprung's disease limited to the rectum and/or sigmoid colon diagnosed on rectal biopsy with established pathological criteria (absence of ganglionic cells +/- hypertrophic extrinsic nerve fibres) (Kapur, Sem Ped Surg 2009),
* Managed successfully with colonic decompressions/irrigations before curative surgery (usually performed 2-3 times a day),
* Uncomplicated form (without enterocolitis and/or diverting colostomy),
* Curative surgery and follow-up in one of the included centres,
* With consent of the 2 parents or legal(s) representative(s),
* Absence of severe or lethal associated malformations,
* Affiliation with the French social security system.

Exclusion Criteria:

* - Long segment Hirschsprung's disease prior to the junction between the left colon and the sigmoid colon,
* Hirschsprung's disease not managed successfully with colonic decompressions/irrigations and requiring a diverting colostomy before the curative surgery,
* Hirschsprung-associated enterocolitis occurring before the randomization,
* Severe or lethal associated malformation, including Down syndrome,
* Intestinal associated malformations (intestinal atresia, gastroschisis, omphalocele, intestinal malrotation and volvulus),
* Any pathological condition that can modify intestinal motility or intestinal transit time (cystic fibrosis, hypothyroidism),
* Refusal of parent(s) or legal representative(s).
* Patients under curatorship or tutorship

Ages: 7 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2019-01-02 (Estimated); Primary Completion 2024-01-02 (Estimated); Study Completion 2024-07-02 (Estimated)

PRIMARY OUTCOMES:
The time to recovery of bowel function after the curative surgery. A 25% decrease of the time to recovery of bowel function in the experimental group as compared to the control group will be considered as clinically effective. | 5 YEARS
  The recovery of bowel function is defined as follows:
  * Tolerance of 2 feeds at full ration (as before surgery, breast-feeding or bottle-feeding),
  * And passing stools.
  The time to recovery of bowel function will be measured in hours from the end of the curative surgery.

SECONDARY OUTCOMES:
The red carmin total transit time will be measured before the surgery | 5 YEARS
  After randomisation (and before the first butyrate enema) Before the curative surgery
The postoperative medium/long-term efficacy of butyrate enemas | 5 YEARS
  Postoperative functional intestinal obstructive symptoms evaluated at each medical appointment The stool consistency evaluated using the validated 'Amsterdam' infant stool form scale at each medical appointment.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France